CLINICAL TRIAL: NCT02625571
Title: Development and Pilot Testing of a Treatment for Children With Sexual Behavior Problems
Brief Title: Tx for Child Sexual Behavior Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Brian Allen, Assistant Professor of Pediatrics, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002942
Record Dates: First submitted 2015-12-02; First posted 2015-12-09 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Phase-based treatment of sexual behavior problems of children

INTERVENTIONS:
Behavioral: Phase-based treatment of sexual behavior problems of children

SUMMARY:
A significant minority of children (ages 5-12) display problematic sexual behavior and the persistence of this behavior is oftentimes as stable as other child behavior problems, such as aggression and defiance. Unfortunately, the only tested intervention protocols for these concerns utilize a group treatment modality that is not feasible in most community treatment settings. This project will define and pilot test an intervention for child sexual behavior problems that is applicable in most settings and can be easily disseminated as a first step toward validation in larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* A caregiver is willing to participate in treatment
* A clinically significant T-score on the Child Sexual Behavior Inventory
* Child is between the ages of 5 and 12, inclusive

Exclusion Criteria:

* Child and/or caregiver IQ below 70
* Active child and/or caregiver psychosis or suicidal/homicidal ideation
* Active substance use problems of the caregiver

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No details to provide. All recruited participants were enrolled.
Groups:
- Intervention: Phase-based treatment of sexual behavior problems of children
Period: Overall Study
Arm/Group | Intervention
Started | 13
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 8 [5 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/European descent | 4
  Non-White/European descent | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Child Sexual Behavior on the Child Sexual Behavior Inventory (CSBI)
Description: Total raw score of the CSBI (potential range = 0-138). Higher scores indicate a greater number and frequency of reported problematic sexual behavior.
Time Frame: 4-6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
Scores on a scale
  Pre-Treatment | 28.8 (17.0)
  Post-Treatment | 18.1 (19.2)

2. Secondary Outcome: Child Sexual Concerns on the Trauma Symptom Checklist for Young Children (TSCYC)
Description: The sexual concerns subscale on the TSCYC provides another metric of sexual behaviors of children. Scaore are reported in T-score, which have a mean of 50 and a standard deviation of 10. A score of 65-70 typically indicates a borderline or sub-syndromal level of concern, while a score of 70 or above indicates clinically significant concern. As such, a higher score indicates greater concern. While there is technically no limit for calculating minimum and maximum values, the reported range of scores is typically between 40 and 100.
Time Frame: 4-6 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
Score on a scale
  Pre-treatment | 80.0 (17.7)
  Post-treatment | 69.6 (26.2)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT02625571/Prot_SAP_000.pdf